CLINICAL TRIAL: NCT00127972
Title: A Retrospective Study to Compare the 3-Year Antiviral Efficacy of Nevirapine and Efavirenz in Combination With D4t and 3tc in 2NN Patients and of Trizivir Versus Trizivir Plus Nevirapine in CHARM Patients
Brief Title: 2NN & CHARM Long-Term Follow-up Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: International Antiviral Therapy Evaluation Center (Other)
Collaborators: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: 04IAT0035
Record Dates: First submitted 2005-08-08; First posted 2005-08-09 (Estimated); Last update posted 2007-04-30 (Estimated); Status verified 2007-04

CONDITIONS: HIV Infections
Keywords: nevirapine; efavirenz; hiv-1; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Stavudine; Lamivudine; Nevirapine; efavirenz; abacavir, lamivudine, and zidovudine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: stavudine
Drug: lamivudine
Drug: nevirapine
Drug: efavirenz
Drug: trizivir

SUMMARY:
It is desirable to obtain extended follow up data on subjects who participated in the 2NN study and the CHARM study in order to see if the beneficial effect of using nevirapine continues up to 144 weeks of treatment.

DETAILED DESCRIPTION:
The 2NN study has been completed, the first large randomised trial comparing the efficacy and safety of ART containing two nucleoside analogue reverse transcriptase inhibitors (nRTI: d4T+3TC) and either NVP-od, NVP-bd, EFV or the combination of NVP+EFV in the treatment of chronically HIV-1 infected ART naive patients. Data from this randomized study show no significant differences in response to treatment, and virologic and immunologic efficacy in the single NNRTI arms NVP-od, NVP-bd and EFV. This contrasts with previous cohort studies, which showed a relative hazard in virologic or treatment failure of more than two for those starting with NVP compared to those starting with EFV.

Despite the results of the 2NN study, question remains whether the comparability of NVP and EFV is maintained over a longer period of follow-up. Therefore, this study is designed to assess the durability of the efficacy of the regimens used in the 2NN study.

In the initial CHARM study, the effect of adding nevirapine and/or hydrea to a triple NRTI regimen (trizivir i.e. abacavir, lamivudine and zidovudine) in terms of efficacy and tolerability was investigated in anti retroviral naïve patients. The primary endpoint was treatment failure and follow up was 72 weeks. A total of 229 patients were included. The use of hydrea was prematurely stopped because adding hydrea significantly contributed to treatment failure through enhancement of the toxicities associated with its use. Subjects in the nevirapine group reached a plasma HIV-1 RNA level < 50 copies/ml quicker (log rank test p = 0.011). In addition, in an as treated analysis only 16.2% of subjects adding nevirapine versus 39.5% adding no nevirapine reached the primary endpoint (p=0.027). These results resemble the findings in the ACTG A5059 study. The trizivir arm of this ACTG study was stopped, because anti-retroviral naïve subjects randomized to receive trizivir experienced virological failure earlier and more frequent than subjects who were randomized to receive either of the two other treatment regimens being evaluated in that study. The two other treatment regimens were:

1. a combination of zidovudine plus lamivudine plus efavirenz and
2. trizivir plus efavirenz.

It is desirable to obtain extended follow up data on subjects who participated in the CHARM study in order to see if the beneficial effect of adding nevirapine to trizivir continues or even increases after 72 weeks of treatment.

In addition to this main objective, another important issue regards the known association between the use of nevirapine and the occurrence of certain untoward effects, including the development of rash, clinical hepatitis and a hypersensitivity syndrome which usually presents with rash, elevated alanine aminotransferase and/or aspartate aminotransferase, eosinophilia and a host of other constitutional symptoms. The possibility that a metabolite of nevirapine might be responsible for one or the other of these events has been evaluated but could not be confirmed. Data is equivocal on whether nevirapine levels themselves are associated with these events, probably because of "noise" in the retrospective analyses that was used. Animal models would suggest, though, that supratherapeutic nevirapine levels are associated with these events. It seems reasonable to assume that there is a sub-population of people at risk for all of these events (especially hypersensitivity) based on their genetic make-up in that it is known that many patients easily tolerate significantly elevated levels of nevirapine while others may get these side effects with relatively normal levels.

To facilitate the safe administration of nevirapine to patients, this study also aims to identify a gene or genes closely associated with these events, and from that a phenotype associated with that genotype which is at increased risk.

ELIGIBILITY:
Inclusion Criteria:

* Participation in the original 2NN or CHARM study

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 763 (Actual)
Dates: Start 2004-02; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
To determine whether the number of patients with treatment failure after 144 weeks of follow-up is different between study arms

SECONDARY OUTCOMES:
To determine whether the percentage of patients with treatment failure after 144 weeks of follow-up is different between the treatment arms
To determine whether the percentage of patients with virologic failure after 144 weeks of follow-up is different between the treatment arms

CONTACTS AND LOCATIONS:
Overall Officials: Joep MA Lange, MD PhD, Study Chair — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Mark Bloch, MD, Principal Investigator — Holdsworth House General Practice
Locations (1):
- Holdsworth House Medical Practice, Darlinghurst, Australia